CLINICAL TRIAL: NCT01932125
Title: An Indian Multicentric, Open Label, Prospective Phase 4 Study of Bevacizumab in the Front Line Management of Advanced/Metastatic Epithelial Ovarian Cancer, Fallopian Tube Cancer or Primary Peritoneal Cancer in Real-life Clinical Practice
Brief Title: An Interventional Study of Avastin (Bevacizumab) in Patients With Advanced/Metastatic Epithelial Ovarian Cancer, Fallopian Tube Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28446
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Experimental)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Participants will receive five cycles of bevacizumab 15 mg/kg concurrently with six cycles of the standard chemotherapy every three weeks (q3w), followed by extended cycles of bevacizumab 15 mg/kg q3w as a single agent for additional 16 cycles. A total of 21 cycles of bevacizumab will be administered in this study.
  Other Names: Avastin

SUMMARY:
This multicenter prospective study will evaluate the safety and efficacy of Avastin (bevacizumab) in routine clinical practice in patients with advanced/metastatic epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer. Data will be collected from eligible patients until death, withdrawal of consent, loss to follow-up, or study closure.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed to receive bevacizumab or already ongoing on treatment with bevacizumab for advanced/metastatic ovarian cancer, fallopian tube cancer or primary peritoneal cancer (FIGO Stage IIIb, IIIc and IV) according to routine clinical practice

Exclusion Criteria:

* Not eligible for treatment with bevacizumab according to the local prescribing information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | up to approximately 1.5 years

SECONDARY OUTCOMES:
Progression-free survival | up to approximately 1.5 years
Overall survival | up to approximately 1.5 years
Overall response rate (complete response + partial response) | up to approximately 1.5 years
Clinical benefit rate (complete response + partial response + stable disease) | up to approximately 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- India (13):
  - Manipal Hospital, Bangalore, Karnataka
  - HealthCare Global Enterprises Limited, Banglore, Karnataka
  - Marthwada Regional Cancer Center & Research Institute, Aurangabad, Maharashtra
  - MOC Cancer Care & Research Centre, Mumbai, Maharashtra
  - HCG NCHRI Cancer Center, Nagpur, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Apex Wellness Hospital, Nashik, Maharashtra
  - Grant Medical Foundation, Ruby Hall Clinic, Pune, Maharashtra
  - Jehangir Clinical Development Centre Pvt. Ltd, Pune, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Rajiv Gandhi Cancer Inst.&Research Center, New Delhi, National Capital Territory of Delhi
  - Peerless Hospitex Hospital and Research Center Ltd., Kolkata, West Bengal
  - MAX Balaji Hospital, Delhi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials Registry - India — http://ctri.nic.in/Clinicaltrials/pmaindet2.php?trialid=5825&EncHid=&userName=Bevacizumab